CLINICAL TRIAL: NCT01847053
Title: A Single-Center, Partial Double-Blind, Randomized, Four-Treatment Crossover Bioavailability Study of Cinnamon in Healthy Subjects
Brief Title: Bioavailability Study of Cinnamon in Healthy Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: McCormick and Company, Inc. (Industry)
Collaborators: Appalachian State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: PRV-1208; MKC-ct01-cn (Other: McCormick)
Record Dates: First submitted 2013-05-01; First posted 2013-05-06 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2015-04

CONDITIONS: Healthy Males
Keywords: Cinnamon; Bioavailability; Glucose; Proanthocyanidins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Oatmeal control (Placebo Comparator): Oatmeal control, around 70g; without cinnamon
  Interventions: Other: Oatmeal
- Ground cinnamon, 3g (Active Comparator): 3 g ground cinnamon in Oatmeal (~70 g)
  Interventions: Other: cinnamon
- Cinnamon extract, 3 g (Active Comparator): 3 g cinnamon extract in Oatmeal (~70 g)
  Interventions: Other: cinnamon
- Cinnamon extract, 6 g (Active Comparator): 6 g cinnamon extract in Oatmeal (~70 g)
  Interventions: Other: cinnamon

INTERVENTIONS:
Other: cinnamon — Intervention will be both ground cinnamon and cinnamon extract.
  Arms: Cinnamon extract, 3 g; Cinnamon extract, 6 g; Ground cinnamon, 3g
Other: Oatmeal — Oatmeal control, around 70g; without cinnamon
  Arms: Oatmeal control

SUMMARY:
A partial double-blind, randomized, placebo-controlled, 4-treatment crossover study design will be used to evaluate bioavailability of various forms of cinnamon and to determine the effects of 3 and 6 g of cinnamon added to instant oatmeal on blood glucose levels in 8 healthy subjects. In the extended dose response study, three subjects will continue the study and be offered 5 day consecutive feedings of 9 g cinnamon extract and on Day 6, and blood samples would be collected over 6 hours after a single morning dose. Urinary samples would be collected upon to 48 hours.

DETAILED DESCRIPTION:
Objective:

The objective of this trial is to evaluate the bioavailability of selected procyanidin derived metabolites from various forms of cinnamon.

Study Products:

Core Study

* Control: Oatmeal (~70 g) without cinnamon
* Active A: Oatmeal (~70 g) with 3 g ground cinnamon
* Active B: Oatmeal (~70 g) with 3 g cinnamon extract
* Active C: Oatmeal (~70 g) with 6 g cinnamon extract

Extension Study

•9 g cinnamon extract in capsule form (unblinded) The 9 g/d cinnamon extract will be consumed by subjects on days 22 through 26. At visit 6 (day 27), subjects will return to the clinic for the test day. The cinnamon extract capsule (9 g) will be consumed with an oatmeal (70 g) breakfast.

Subjects:

Subjects will be healthy men 18 - 40 years of age (inclusive), each with a body mass index (BMI) 25.00-29.99 kg/m2.

Outcome Variables:

Primary Outcome Variable The primary outcome variables will be the area under the curve (AUC) from 0 to 360 min for plasma procyanidin-derived metabolites, where t=0 min is the start of study product consumption.

Secondary Outcome Variables

Secondary outcome variables will include the assessment of:

* The maximum concentration (Cmax) and time to reach peak concentration (Tmax) for plasma procyanidin-derived metabolites, as well as the net incremental AUC values to account for possible non-zero pre-load values.
* The effect of a single dose of cinnamon on the metabolic profile using an untargeted metabolomics analysis on both plasma and urine specimens.
* The effect of a single dose of cinnamon on plasma glucose and insulin.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a healthy male, 18 - 40 years of age, inclusive.
2. Subject has a body mass index (BMI) 25.00-29.99 kg/m2
3. Subject is willing to discontinue dietary supplement use for 2 weeks prior to the first test visit
4. Subject is willing to avoid foods high in procyanidins for 2 d prior to the first test visit (visit 2, day 0) and throughout the trial.
5. Subject does not smoke and has no plans to change smoking habits during the study period.
6. Subject has a score of 7 to 10 on the Vein Access Scale at visit 1 (day -3;
7. Subject is judged by the Investigator to be in general good health on the basis of physical examination and medical history.
8. Subject understands the study procedures and signs forms providing informed consent to participate and authorization for release of relevant protected health information to the study Investigators.

Exclusion Criteria:

1. Subject has a history or presence of a gastrointestinal condition that could potentially interfere with absorption of the study product (e.g. inflammatory bowel syndrome, celiac disease, history of gastric bypass surgery).
2. Subject has a history or presence of clinically important endocrine (including type 1 or 2 diabetes mellitus), cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, renal, hepatic, pancreatic, biliary or neurologic disorders that, in the opinion of the Investigator, could interfere with the interpretation of the study results.
3. Subject has a history or presence of cancer in the prior two years, except for non-melanoma skin cancer.
4. Subject has a current infection at visit 1 (day -3) or subject has an active infection or use of antibiotics within 5 d of any test visit (visits 2 through 5; days 0 through 21) and extension visit [visit 6 (day 27); for the subset of subjects participating in the extension]. For those with an active infection and/or using antibiotics, subjects must wait at least 5 d after the infection resolves or antibiotic use is complete to participate in a test visit.
5. Subject has consumed alcoholic beverages within 24 h of any test day (visits 2 through 5; days 0 through 21) and the extension visit [visit 6 (day 27); for the subset of subjects participating in the extension].
6. Subject has used any over-the-counter or prescription medications within 4 weeks of visit 1 (day -3)
7. Subject has a history of any major trauma or major surgical event within 3 months of visit 1 (day -3).
8. Subject has hypertension (systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg) at visit 1 (day -3).
9. Subject has a history of allergy or sensitivity to any of the components of the study products, standard meal/snack or liquid meal.
10. Subject has been exposed to any non-registered drug product within 30 d prior to visit 1 (day -3).
11. Subject has a current or recent history (past 12 months of visit 1) or strong potential for drug or alcohol abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor).
12. Individual has a condition the Investigator believes would interfere with his ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome variables will be the area under the curve (AUC) from 0 to 360 min for plasma procyanidin-derived metabolites. | up to 12 months

SECONDARY OUTCOMES:
•The effect of a single dose of cinnamon on the metabolic profile. | up to 12 months
  The metabolites and metabolic profile will be analyzed using targeted and untargeted metabolomics analysis on both plasma and urine specimens.
•The effect of a single dose of cinnamon on plasma glucose and insulin. | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maki, PhD, Principal Investigator — Biofortis Clinical Research, Inc.
Locations (1):
- Biofortis Clinical Research, Addison, Illinois, United States